CLINICAL TRIAL: NCT04043819
Title: Evaluation of Safety and Exploratory Efficacy of PSC-01, an Autologous Adipose-derived Stromal Vascular Fraction Cell Therapy Product for the Treatment of Knee Osteoarthritis
Brief Title: Evaluation of Safety and Exploratory Efficacy of an Autologous Adipose-derived Cell Therapy Product for Treatment of Single Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Personalized Stem Cells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-CP-001
Record Dates: First submitted 2019-07-23; First posted 2019-08-02 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
Keywords: cellular therapy; stromal vascular fraction; SVF; KOOS; autologous; mesenchymal stem cell; MSC; knee; osteoarthritis; adipose-derived mesenchymal stem cells; Ad-MSC; intraarticular
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PSC-01 (Experimental): All study participants will receive intraarticular injection of the investigational biological product, PSC-01.
  Interventions: Drug: PSC-01

INTERVENTIONS:
Drug: PSC-01 — PSC-01 is a form of autologous cellular therapy resulting from the enzymatic processing of lipoaspirate to yield adipose-derived stromal vascular fraction cells.

SUMMARY:
The objective of this clinical study is to evaluate the safety of an intraarticular injection of an investigational biologic product (IBP), PSC-01, the patient's own adipose-derived stromal vascular fraction cells (SVF) extracted from a lipoaspirate sample, to treat the pain of osteoarthritis in a single knee. The secondary objective is to get initial data on efficacy of the PSC-01.

ELIGIBILITY:
Inclusion Criteria:

* If a woman of childbearing potential, the study participant must not be pregnant at the time of consent and must take contraceptive measures to prevent a pregnancy while actively participating in the study
* The study participant may be of any gender or ethnic background.
* Must experience knee pain at least weekly for at least 3 months.
* Must have failed a minimum of 6 weeks of first line, conservative therapy
* Demonstrated clinical and radiographic evidence of OA diagnosis
* Grade 2, 3, or 4 Kellgren-Lawrence score in one knee.
* Normal or within protocol approved limits of laboratory blood and urinalysis tests
* Must be suitable for cellular therapy per the Investigator's opinion
* Must be suitable for liposuction per the Investigator's opinion
* Must possess the cognitive ability to understand the investigational nature of this clinical trial and voluntarily provide consent for study participation

Exclusion Criteria:

* Evidence of OA in the contralateral knee with a Kellgren-Lawrence score greater than 2
* If a woman of child-bearing potential, the study participant must not be pregnant or attempt to become pregnant while actively taking part in the study.
* Steroid injection in either knee within 60 days of providing informed consent
* The subject must not be diagnosed with any of the following diseases at the time of consent:

  * Osteonecrosis
  * Active autoimmune disease
  * Serious cardiac condition
  * Psychotic Diseases
  * Epilepsy
  * Uncontrolled diabetes
* Prescribed immunosuppressive therapy at the time of consent
* Evidence of cancer at the time of consent
* History of alcohol or substance abuse
* Regular smoker at the time of consent
* Received experimental medication or participated in another clinical study within 60 days of providing informed consent
* Concurrent diseases or circumstances that the Investigator judges to be a potential risk to patient health or a confounding variable in the assessment of study endpoints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 3-4 months
  The primary outcome measure of this study is to evaluate the safety of the investigational biological product, PSC-01.Safety will be assessed as the number of treatment-related adverse events as assessed by CTCAE v5.0. Adverse events will be assessed by physical examination, patient-reported health status, clinical pathology evaluations (cbc, chemistry, and urinalysis), and post-procedure clinical observations through the 84-day study period with post-treatment follow-up at 6 and 12 months.

SECONDARY OUTCOMES:
Changes in KOOS Measurement | 3-4 months
  The secondary outcome measure of this study is to obtain initial data on the efficacy of PSC-01 on treating knee osteoarthritis. The efficacy primary outcome will be assessed using the KOOS knee survey with the five relevant subcategories of pain, symptoms, average daily living, sport/recreation, and quality of life measured at baseline, day 42 and day 84.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - San Diego Orthobiologics Medical Group, Carlsbad, California
  - Grossmont Orthopedic Medical Group, La Mesa, California
  - Synergy Orthopedic Specialists Medical Group, San Diego, California
  - The Orthohealing Center, Santa Monica, California
  - Cellular Orthopedics, Des Plaines, Illinois
  - New Jersey Regenerative Institute, Cedar Knolls, New Jersey
  - RestorePDX, Beaverton, Oregon

REFERENCES:
- [Derived] Rogers CJ, Harman R, Sheinkop MB, Hanson P, Ambach MA, David T, Desai R, Sampson S, Aufierro D, Bowen J, Malanga G. Clinical Evaluation of Safety and Efficacy of a Central Current Good Manufacturing Practices Laboratory Produced Autologous Adipose-Derived Stromal Vascular Fraction Cell Therapy Product for the Treatment of Knee Osteoarthritis. Stem Cells Dev. 2024 Apr;33(7-8):168-176. doi: 10.1089/scd.2024.0008. PMID 38386505